CLINICAL TRIAL: NCT00613587
Title: Effect of Roflumilast In-Vitro on Basophil Histamine, Leukotriene, IL-4 and IL13-release.
Brief Title: Roflumilast In-Vitro Basophil Release
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: RGT2007
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-09

CONDITIONS: Allergy; Asthma
Keywords: Interleukin 13; Interleukin 4; Leukotrienes; Basophil Histamine Release
MeSH Terms: conditions — Hypersensitivity; Asthma; Rhinitis, Allergic

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Polymorphal Blood Mononuclar Cells will be stimulated to release various cytokines. The supernatant of the stimulations will be stored for batched analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is looking for allergic asthmatics. Lung and allergy testing will be done to verify. If qualified, blood will be drawn for laboratory studies.

DETAILED DESCRIPTION:
Non-smoking allergic asthmatics will be verified using pulmonary function, skin prick testing, exhaled nitric oxide and serum IgE. If qualified, blood will be drawn, treated with study medication and then stimulated with the allergen to which the subject is allergic. Mediators including Histamine, IL-13, IL-4, and leukotrienes will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and above Allergic Asthma Serum IgE greater than 30iu/ml Exhaled Nitric Oxide greater than 17ppb

Exclusion Criteria:

* smoking history

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Allergic Asthma, non-smoker
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Townley, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States